CLINICAL TRIAL: NCT04558853
Title: A Safety Study of CellProtect, an Autologous ex Vivo Expanded and Activated Natural Killer (NK) Cell Product, in Patients With Multiple Myeloma
Brief Title: Clinical Study of Autologous Natural Killer Cells in Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Hareth Nahi, Principal Investigator, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-001
Record Dates: First submitted 2020-09-10; First posted 2020-09-22 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Multiple Myeloma
Keywords: NK cells; Consolidation
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous NK cells (Experimental): The investigation product is a cell suspension based on ex vivo expanded NK cells from patients with MM. The treatment is strictly autologous. The IP is given as three infusions with escalating doses.
  Mode of administration Intravenous infusions. Dose levels
  * First infusion; 5x10^6 cells/kg body weight
  * Second infusion; 50x10^6 cells/kg body weight
  * Third infusion; 100x10^6 cells/kg body weight
  Interventions: Drug: autologous NK cells

INTERVENTIONS:
Drug: autologous NK cells — Autologous ex vivo expanded and activated NK cells

SUMMARY:
Multiple Myeloma (MM) is a lethal disease and at present no available treatment method seems to prevent the disease from progressing or relapsing in the long term. NK cells have a relatively high cytotoxic capacity and an anti tumour effect, suggesting a potential as a treatment of MM.This is a phase I, first-in-human, therapeutic exploratory study, where no benefits for the patients can be guaranteed. However, the theoretical implication is that the infused cells may have a positive antitumour effect for the participating individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Above 18 years of age
3. MM diagnosis (stage I-III according to the International Staging System)
4. Eligible for, and willing to undergo, high dose chemotherapy and ASCT
5. Measurable monoclonal immunoglobulins
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
7. Life expectancy of at least three months

Exclusion Criteria:

1. Non-secretory MM
2. Malignancy, other than MM, treated with chemotherapy or radiation within the past six months
3. Blood donation or other significant blood loss within three months from screening
4. Any physical condition or laboratory results that contraindicate a blood donation to be performed within four weeks from screening
5. Any physical condition or laboratory results that require the chemotherapy to start before there is available slot for blood donation
6. Known or suspected allergic reactions to any ingredient of the IP
7. Diagnosis or indication of any active autoimmune disease, such as Rheumatoid Arthritis, Inflammatory Bowel Disease, Systemic Lupus Erythematosis or Multiple Sclerosis
8. Uncontrolled or severe cardiovascular disease, such as myocardial infarction within six months from screening, heart failure (class III or IV according to New York Heart Association), uncontrolled angina, clinically significant pericardial disease or cardiac amyloidosis
9. Poorly controlled hypertension
10. Poorly controlled Diabetes Mellitus, type I or II
11. Diagnosis or indication of any clinically relevant renal disease
12. Diagnosis or indication of any clinically relevant hepatic disease
13. Ongoing infection that is considered chronic
14. Known or suspected drug or alcohol abuse, within 12 months from screening
15. Pregnant, trying to become pregnant, or nursing
16. Lack of, or unreliable contraceptive method, as judged by the Investigator
17. Medical history or any abnormal physical finding that is clinically relevant and could interfere with the safety or objectives of the study, as judged by the Investigator
18. Lack of suitability for participation in the trial, for any reason, as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From first dose of study treatment up until six months from last infusion.
  Assessment of treatment-emergent adverse events/serious adverse events (TEAEs/SEAS)(including IARS). TEAEs are defined as AEs that develop, worsen (according to the Investigators opinion), or bedome serious during the treatment period.

SECONDARY OUTCOMES:
Changes on serum monoclonal immunoglobulin levels as a marker of efficacy | From date of screening through study completion, up until six months from last infusion
  Changes in absolute and relative levels of laboratory parameters
Changes on urine monoclonal immunoglobulin levels as a marker of efficacy | From date of screening through study completion, up until six months from last infusion
  Changes in absolute and relative levels of laboratory parameters
Changes on serum free light chain levels as a marker of efficacy | From date of screening through study completion, up until six months from last infusion
  Changes in absolute and relative levels of laboratory parameters
Effect of CellProtect on plasma cell fraction in bone marrow | From date of screening up until one month from last infusion
  Changes in bone marrow clonal plasma cells
Response assessment as defined by the International Myeloma Working Group uniform response criteria | From date of screening up until six months from last infusion
  Evaluation of response criteria, i.e. minimal response, partial response, very good partial response and complete response as assessed by International Myeloma Working Group uniform response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Hareth Nahi, M.D., Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No